CLINICAL TRIAL: NCT01530399
Title: A Phase II, Double-blind, Parallel Group, Dose-selection Study to Compare Antifibrinolytic MDCO-2010 vs. Placebo and Tranexamic Acid in Reducing Blood Loss in Patients Undergoing Primary Cardiac Surgery
Brief Title: Phase II Study to Compare MDCO-2010 vs Placebo and Tranexamic Acid in Patients Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TMC-MDC-11-01
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Results first posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — 4-(2'-hydroxy-3'-methylbut-3'-enyloxy)-8H-(1,3)dioxolo(4,5-h)chromen-8-one; 3-(4'-methoxybenzyl)-7,8-methylenedioxychroman-4-one; Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MDCO 1 (Experimental): MDCO-2010: load 15 μg/kg; infusion 30 μg/kg/h; CPB prime 0.11 μg/mL priming volume
  Interventions: Drug: MDCO 1
- MDCO 2 (Experimental): MDCO-2010: load 30 μg/kg; infusion 60 μg/kg/h; CPB prime 0.22 μg/mL priming volume
  Interventions: Drug: MDCO 2
- MDCO 3 (Experimental): MDCO-2010: load 60 μg/kg ; infusion 120 μg/kg/h; CPB prime 0.44 μg/mL priming volume
  Interventions: Drug: MDCO 3
- MDCO 4 (Experimental): MDCO-2010: load 90 μg/kg; infusion 180 μg/kg/h; CPB prime 0.65 μg/mL priming volume
  Interventions: Drug: MDCO 4
- Saline (Placebo Comparator): Commercially available saline (0.9% NaCl solution)
  Interventions: Drug: Tranexamic Acid
- Tranexamic acid (Active Comparator): Tranexamic acid: 12 mg/kg loading dose; 5 mg/kg/h infusion; 0.556 mg/mL CPB priming
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: MDCO 1 — MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 1: load 15 μg/kg; infusion 30 μg/kg/h; CPB prime 0.11 μg/mL priming volume
  Other Names: MDCO-2010
  Arms: MDCO 1
Drug: MDCO 2 — MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 2: load 30 μg/kg; infusion 60 μg/kg/h; CPB prime 0.22 μg/mL priming volume
  Other Names: MDCO-2010
  Arms: MDCO 2
Drug: MDCO 3 — MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 3: load 60 μg/kg ; infusion 120 μg/kg/h; CPB prime 0.44 μg/mL priming volume
  Other Names: MDCO-2010
  Arms: MDCO 3
Drug: MDCO 4 — MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 4: load 90 μg/kg; infusion 180 μg/kg/h; CPB prime 0.65 μg/mL priming volume
  Other Names: MDCO-2010
  Arms: MDCO 4
Drug: Tranexamic Acid — Tranexamic acid will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with tranexamic acid. The flow rates will be the same as for MDCO-2010.
  Other Names: TXA
  Arms: Saline
Drug: Saline — A loading dose of saline will be followed by a continuous infusion of saline until sternal closure. In addition, the CPB reservoir will be primed with saline. The flow rates will be the same as for MDCO-2010.
  Other Names: NaCl 0.9%
  Arms: Tranexamic acid

SUMMARY:
The objective of this study is to determine the dose response relationship regarding blood loss, PK, PD and clinical outcomes of MDCO-2010 in comparison to placebo and tranexamic acid in patients undergoing primary cardiac surgery with cardiopulmonary bypass. The aim of the study is to define minimally effective dose of MDCO-2010.

DETAILED DESCRIPTION:
This was a two-stage, double-blind, randomized, parallel-group, multicenter Phase II dose-selection study to compare antifibrinolytic MDCO-2010 vs tranexamic acid and placebo in reducing blood loss.

This study was designed to examine a broad range of doses to fully characterize the dose-response relationship between MDCO-2010 dose, plasma PK, PD, and clinical effects.

In Stage 1, 90 patients were to be enrolled into one of six treatment groups with 15 patients per group: four groups were to receive MDCO-2010, one group was to receive tranexamic acid, and one group was to receive placebo. Stage 2 was to be an expansion of Stage 1.

The study was terminated after 49 patients were enrolled into Stage 1.

ELIGIBILITY:
Inclusion Criteria:

* For Stage 1: Planned primary isolated CABG surgery
* For Stage 2: Planned primary isolated CABG surgery, OR Planned primary combined CABG and aortic valve replacement surgery
* Men, aged 18 to 85 years, or Women, aged 18 to 85 years, either of postmenopausal status, defined as ≥1 year since last menstrual period AND if less than 65 years old with a negative pre-operative pregnancy test within 24 hours of surgery OR with medical history of hysterectomy or bilateral oophorectomy
* Written informed consent

Exclusion Criteria:

* Off-pump surgery or hybrid procedures
* Patients undergoing repeat sternotomy
* Planned deep hypothermic circulatory arrest (<28°C)
* Known allergy, sensitivity, or contraindications to tranexamic acid
* Epileptiform disorders, history of seizure activity, or anticonvulsive medication
* Administration of clopidogrel, ticagrelor or ticlopidine within 5 days prior to surgery or prasugrel within 7 days prior to surgery.
* Administration of low molecular weight heparin, glycoprotein IIb/IIIa inhibitors, or fondaparinux within 12 hours prior to surgery
* Known history of coronary stent thrombosis within the last three months
* History of stroke or transient ischemic attack within 3 months prior to surgery
* History of deep venous thrombosis or pulmonary embolism
* LVEF ≤35% or Grade III or IV
* Body mass index <20 or >35
* Known active gastrointestinal (GI) or other non-catheterization bleeding within 7 days prior to surgery
* Preoperative coagulation abnormalities defined as:
* Platelet count <100,000/L or >350,000/L, or
* International normalized ration (INR) >1.5, or
* Hematocrit <36%, or
* aPTT >1.5 x ULN
* Major surgical procedures within 30 days prior to surgery
* Patient inability or refusal to receive donor blood products if necessary
* Creatinine >2 mg/dL or estimated glomerular filtration rate (eGFR) (calculated using Modification of Diet in Renal Disease [MDRD] equation <30 mL/min)
* Known heparin-induced thrombocytopenia type II
* Known history of thrombophilia, such as AT-III, Protein C or Protein S deficiency, Factor V Leiden, anti-phospholipid syndrome
* Active liver disease defined as any known current infectious, neoplastic or metabolic pathology of the liver OR ALT or AST elevation >2x ULN or total bilirubin elevation >1.5x ULN at Screening
* Any condition requiring ongoing chronic immunosuppressive medication
* Malignancy within 5 years prior to surgery
* Receipt of an investigational drug or device within 60 days prior to surgery Any other condition which, in the opinion of the Principal Investigator, would put the subject at increased risk from participating in the study or otherwise prevent a patient"s participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Englberger, PD DR. med, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (5):
- Germany (4):
  - Charité Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universität Heidelberg, Heidelberg
  - Universität Leipzig - Herzzentrum, Leipzig
- University Hospital/Inselspital Bern, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- MDCO 1: MDCO-2010 Dose 1: MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 1: load 15 μg/kg; infusion 30 μg/kg/h; CPB prime 0.11 μg/mL priming volume
- MDCO 2: MDCO-2010 Dose 2: MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 2: load 30 μg/kg; infusion 60 μg/kg/h; CPB prime 0.22 μg/mL priming volume
- MDCO 3: MDCO-2010 Dose 3: MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 3: load 60 μg/kg ; infusion 120 μg/kg/h; CPB prime 0.44 μg/mL priming volume
- MDCO 4: MDCO-2010 Dose 4: MDCO-2010 will be administered as a loading dose followed by a continuous infusion until sternal closure. In addition, the CPB reservoir will be primed with MDCO-2010. MDCO 4: load 90 μg/kg; infusion 180 μg/kg/h; CPB prime 0.65 μg/mL priming volume
Period: Overall Study
Arm/Group | MDCO 1 | MDCO 2 | MDCO 3 | MDCO 4 | Saline | Tranexamic Acid
Started | 8 | 10 | 8 | 10 | 6 | 7
Completed | 7 | 8 | 7 | 10 | 6 | 6
Not Completed | 1 | 2 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MDCO 1 | MDCO 2 | MDCO 3 | MDCO 4 | Saline | Tranexamic Acid | Total
Number analyzed (Participants) | 8 | 10 | 8 | 10 | 6 | 7 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [64 to 75] | 70 [57 to 73] | 66 [60 to 79] | 73 [68 to 73] | 66 [60 to 71] | 58 [52 to 62] | 69 [61 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 2 | 0 | 8
  Male | 7 | 8 | 7 | 8 | 4 | 7 | 41
Region of Enrollment [Number; unit: participants]
  Germany | 6 | 7 | 5 | 7 | 4 | 4 | 33
  Switzerland | 2 | 3 | 3 | 3 | 2 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Chest Tube Drainage at 12 Hours After Surgery
Time Frame: 12 hours post CABG
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | MDCO 1 | MDCO 2 | MDCO 3 | MDCO 4 | Saline | Tranexamic Acid
Number analyzed (Participants) | 7 | 7 | 6 | 10 | 6 | 6
mL | 600 [300 to 970] | 580 [420 to 880] | 480 [350 to 700] | 453 [415 to 645] | 645 [400 to 1040] | 593 [530 to 750]

ADVERSE EVENTS:
Time Frame: 30 (+5) days post treatment
Arm/Group | MDCO 1 | MDCO 2 | MDCO 3 | MDCO 4 | Saline | Tranexamic Acid
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/8 | 1/7 | 2/10 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/7 | 7/8 | 4/7 | 7/10 | 5/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDCO 1 (N=7) | MDCO 2 (N=8) | MDCO 3 (N=7) | MDCO 4 (N=10) | Saline (N=6) | Tranexamic Acid (N=6)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Low cardiac output syndrome (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDCO 1 (N=7) | MDCO 2 (N=8) | MDCO 3 (N=7) | MDCO 4 (N=10) | Saline (N=6) | Tranexamic Acid (N=6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 1 | 2 | 1 | 2
Troponin T increased (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 2 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
AST increased (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0 | 0
AST increased (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After initial multicenter results communications are published, or after 12 months from study closure (whichever occurs first), sponsor can review results communications prior to submission and can embargo submissions for a period of 45 days from the time submitted to the sponsor for review, agreeing to resolve differences of opinion or interpretation through scientific debate. Sponsor can request further delay for an additional 90 days to file any patent applications if deemed necessary